CLINICAL TRIAL: NCT03978195
Title: EMD - A Non-invasive Device for Ventilating the Middle Ear Feasibility Study to Evaluate Efficiency and User Satisfaction
Brief Title: A Non-invasive Device to Remove Fluid From the Middle Ear
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Yuinvent Innovations Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0275-18-MMC (CLEAR OM R1)
Record Dates: First submitted 2019-06-03; First posted 2019-06-07 (Actual); Last update posted 2019-06-07 (Actual); Status verified 2019-06

CONDITIONS: Otitis Media With Effusion
MeSH Terms: conditions — Otitis Media with Effusion | interventions — Middle Ear Ventilation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Treatment (Experimental)
  Interventions: Device: Non-invasive device for middle ear ventilation
- Control (No Intervention)

INTERVENTIONS:
Device: Non-invasive device for middle ear ventilation — Daily use of the device
  Arms: Treatment

SUMMARY:
A feasibility study for evaluating efficacy and satisfaction is treated using a non-invasive device for middle ear ventilation.

The study is designed to test the device's effectiveness by encouraging the evacuation of fluid from the middle ear, aid in hearing improvement, pain relief and assessment of patient satisfaction with the use of the device.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with ear fluids (OME) according to a doctor's examination for at least 4-6 weeks. There is a progressive hearing impairment and a matching tympanum.
* In principle, these children (with OME and hearing impairment) meet the criteria and candidates for the analysis of inserting tubes of incontinence (buttons).

Exclusion Criteria:

* First encounter: acute ear infection or Proper Otoscopy
* Second session: First review: Otoscopy / Timpneometry / Hearing test.
* Parallel treatment: acupuncture - tubes insertion - discontinuation of follow-up - cessation of the experiment initiated by parents

Ages: 4 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2019-07-01 (Estimated); Primary Completion 2021-08-01 (Estimated); Study Completion 2021-11-01 (Estimated)

PRIMARY OUTCOMES:
Middle ear values of Tympanometry | 10 weeks
  Values will be compared to baseline values of Tympanometry
Middle ear ventilation evaluated by otoscopy | 10 weeks
  Otoscopy evaluation of ear ventilation will be compared to baseline values

SECONDARY OUTCOMES:
Auditory test | 10 weeks
  Values will be compared to baseline values of Auditory test

IPD SHARING:
Plan to Share IPD: No